CLINICAL TRIAL: NCT07016789
Title: Cerebral Regional Oxygen Saturation During TAVI: A Prospective Comparison of Balloon-Expandable and Self-Expanding Valves
Brief Title: Cerebral Regional Oxygen Saturation During TAVI - The CROS-TAVI Prospective Registry
Acronym: CROS-TAVI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7257
Record Dates: First submitted 2025-05-29; First posted 2025-06-12 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-04

CONDITIONS: Aortic Stenosis Disease; TAVI(Transcatheter Aortic Valve Implantation); Cerebral Oxygen Saturation; Hemodynamic Changes
Keywords: TAVI; Aortic Valve Stenosis; Cerebral Oxygen Saturation; NIRS; Balloon-Expandable Valve; Self-Expanding Valve
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:1 ratio to receive either a balloon-expandable valve (Group A) or a self-expanding valve (Group B).
  Patients randomized to Group B will undergo a second randomization to receive either:
  an intra-annular SEV (Group B1 - NAVITOR), or a supra-annular SEV (Group B2 - EVOLUT). Patients will be randomized in a 1:1 ratio to receive either a balloon-expandable valve (Group A) or a self-expanding valve (Group B).
  Patients randomized to Group B will undergo a second randomization to receive either:
  an intra-annular SEV (Group B1 - NAVITOR), or a supra-annular SEV (Group B2 - EVOLUT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Balloon-expandable valve (Group A) (Experimental): Participants in this arm will receive a balloon-expandable transcatheter heart valve (SAPIEN platform, Edwards Lifesciences). Cerebral oxygenation will be monitored during the TAVI procedure using NIRS.
  Interventions: Device: Near-infrared spectroscopy monitoring (NIRS) INVOS 5100C
- Self-expanding intra-annular valve (Group B1) (Experimental): Participants in this arm will receive an intra-annular self-expanding valve (NAVITOR, Abbott). Cerebral rSO₂ will be monitored during TAVI using NIRS at predefined timepoints.
  Interventions: Device: Near-infrared spectroscopy monitoring (NIRS) INVOS 5100C
- Self-expanding supra-annular valve (Group B2) (Experimental): Participants in this arm will receive a supra-annular self-expanding valve (EVOLUT, Medtronic). NIRS will be used to monitor cerebral oxygenation throughout the TAVI procedure.
  Interventions: Device: Near-infrared spectroscopy monitoring (NIRS) INVOS 5100C

INTERVENTIONS:
Device: Near-infrared spectroscopy monitoring (NIRS) INVOS 5100C — Continuous bilateral cerebral oxygen saturation monitoring using near-infrared spectroscopy (NIRS) during TAVI. Sensors are placed on the forehead to record rSO₂ values at predefined timepoints. Device used: INVOS 5100C (Medtronic/Covidien).

SUMMARY:
This single-center, non-commercial clinical study investigates how different types of transcatheter aortic valve prostheses affect cerebral oxygen saturation during the procedure (TAVI - Transcatheter Aortic Valve Implantation). The study uses a non-invasive monitoring system (NIRS) to track brain oxygenation (rSO₂) in real time.

The goal is to understand whether balloon-expandable, intra-annular self-expanding, or supra-annular self-expanding valves lead to different levels or patterns of cerebral oxygenation. This may help identify early warning signs for delayed hemodynamic recovery, stroke, or delirium.

Participants will be randomly assigned to receive one of:

A balloon-expandable valve (Group A), or

A self-expanding valve (Group B), with further randomization into:

Group B1: intra-annular valve (NAVITOR)

Group B2: supra-annular valve (EVOLUT)

The procedure, follow-up, and data collection will follow standard clinical practice. No experimental devices or drugs are used. Patients will not undergo any additional risk or burden beyond what is normally expected during TAVI.

The study is being conducted at the Fondazione Policlinico Universitario A. Gemelli IRCCS in Rome, Italy, and aims to enroll 40 patients. No compensation is provided, and participation is voluntary.

DETAILED DESCRIPTION:
This is a prospective, randomized, single-center, interventional clinical study conducted at the Fondazione Policlinico Universitario A. Gemelli IRCCS in Rome, Italy. The study aims to investigate differences in cerebral regional oxygen saturation (rSO₂) during transcatheter aortic valve implantation (TAVI) using different transcatheter heart valve (THV) technologies.

Aortic valve stenosis (AVS) is the most common valvular disease in the elderly, and TAVI has become a widely accepted therapeutic option in high-, intermediate-, and low-risk patients. However, the rapid ventricular pacing, balloon dilatation, and valve deployment involved in TAVI may induce transient cerebral hypoperfusion. This study utilizes near-infrared spectroscopy (NIRS) as a non-invasive method to monitor cerebral oxygenation in real-time during the procedure.

The primary objective is to evaluate the variation in rSO₂ during specific procedural phases and determine whether the type of valve used (balloon-expandable vs. self-expanding) impacts cerebral perfusion. A secondary aim is to identify a potential threshold value of rSO₂ below which prolonged hemodynamic recovery may occur. The study also explores the association between cerebral desaturation and clinical outcomes such as in-hospital mortality, stroke, and postprocedural delirium.

Patients with symptomatic severe aortic stenosis meeting specific inclusion/exclusion criteria will be enrolled and randomized 1:1 to receive:

Group A: A balloon-expandable valve (SAPIEN platform, Edwards Lifesciences)

Group B: A self-expanding valve (SEV)

Patients in Group B will be further randomized to receive:

Group B1: Intra-annular SEV (NAVITOR, Abbott)

Group B2: Supra-annular SEV (EVOLUT, Medtronic)

Cerebral rSO₂ will be monitored bilaterally using INVOS 5100C NIRS sensors placed on the forehead. Measurements will be recorded at six procedural time points: baseline (pre-induction), start of procedure, during pre-dilatation (if performed), at valve deployment, at the lowest rSO₂ during deployment, post-dilatation (if performed), and end of procedure.

Neurocognitive status will be assessed pre-procedure using the Mini-Mental State Examination (MMSE). Postoperative delirium will be monitored using the CAM-ICU and RASS scales. Clinical and procedural data, including rapid ventricular pacing parameters, valve type, and any need for resheathing, will also be recorded.

The primary endpoint is the comparison of mean nadir rSO₂ values between balloon-expandable and self-expanding valve groups. Exploratory analyses will evaluate differences among all three groups (A, B1, B2). Secondary endpoints include in-hospital death, stroke, and delirium incidence.

A total of 40 patients will be enrolled (20 in Group A, 10 in B1, 10 in B2). The study is no-profit, does not involve investigational drugs or unapproved devices, and all THVs used are CE-marked and clinically approved. The protocol has been approved by the local ethics committee (CET Lazio Area 3, ID 7257).

The findings of this study may provide novel insights into the role of cerebral oxygenation monitoring during TAVI and contribute to optimizing valve selection and procedural strategies to improve neurologic and hemodynamic outcomes.

ELIGIBILITY:
Inclusion Criteria:

Signed informed consent prior to any study-specific procedures

Diagnosis of severe degenerative aortic valve stenosis with echocardiographic criteria:

Mean gradient > 40 mm Hg, or

Jet velocity > 4.0 m/s, or

Aortic valve area (AVA) < 0.8 cm² (or AVA index < 0.5 cm²/m²)

Symptomatic aortic stenosis defined as NYHA functional class ≥ II

Exclusion Criteria:

Symptomatic carotid artery disease or indication for carotid revascularization

Cardiogenic shock or inotropic support required prior to the procedure

Active neurodegenerative disease

Contraindications as determined by anesthesiology screening

Age < 18 years

Contraindications to NIRS monitoring

ST-elevation myocardial infarction or cardiogenic shock within 48h before enrollment

Emergency TAVI due to decompensated AV stenosis

Malignancy or comorbidities with life expectancy < 12 months

Inability to comply with the study protocol

Stroke or transient ischemic attack within 6 months

Renal insufficiency (creatinine > 3.0 mg/dL) or dialysis dependency

Severe left ventricular dysfunction (LVEF < 30%)

Significant mixed valvular disease (e.g., severe mitral or tricuspid regurgitation)

Intracardiac mass, thrombus, or vegetation

Chronic corticosteroid use

Participation in another investigational drug or device study

Active bacterial endocarditis or other active infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in cerebral regional oxygen saturation (rSO₂) during transcatheter aortic valve implantation (TAVI) | Intraoperative, from pre-induction to end of TAVI procedure (approximately 60-90 minutes)
  Cerebral rSO₂ will be monitored at six procedural timepoints using NIRS: pre-induction, start of procedure, pre-dilatation (if performed), valve deployment, lowest rSO₂ value during deployment, post-dilatation (if performed), and end of procedure. The primary outcome is the comparison of rSO₂ profiles between patients receiving balloon-expandable valves and those receiving self-expanding valves.

SECONDARY OUTCOMES:
In-hospital all-cause mortality | From procedure to hospital discharge (up to 14 days)
  Number of participants who die from any cause during the index hospitalization after TAVI.
In-hospital stroke incidence | From procedure to hospital discharge (up to 14 days)
  Occurrence of stroke during the hospitalization period, as defined by VARC-3 criteria.
Incidence of postoperative delirium | First 3 days after the procedure or until discharge from ICU
  Delirium will be assessed using CAM-ICU and RASS scales during the first three days post-TAVI or ICU stay.

OTHER OUTCOMES:
Exploratory comparison of cerebral oxygen saturation across all three valve types | Intraoperative, from pre-induction to end of TAVI procedure (approximately 60-90 minutes)
  Exploratory analysis of cerebral rSO₂ trends and nadir values during TAVI among three groups: balloon-expandable (Group A), intra-annular self-expanding (Group B1), and supra-annular self-expanding valves (Group B2). The analysis will investigate whether different valve designs result in different cerebral oxygenation patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Aurigemma, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] VARC-3 WRITING COMMITTEE:; Genereux P, Piazza N, Alu MC, Nazif T, Hahn RT, Pibarot P, Bax JJ, Leipsic JA, Blanke P, Blackstone EH, Finn MT, Kapadia S, Linke A, Mack MJ, Makkar R, Mehran R, Popma JJ, Reardon M, Rodes-Cabau J, Van Mieghem NM, Webb JG, Cohen DJ, Leon MB. Valve Academic Research Consortium 3: Updated Endpoint Definitions for Aortic Valve Clinical Research. J Am Coll Cardiol. 2021 Jun 1;77(21):2717-2746. doi: 10.1016/j.jacc.2021.02.038. Epub 2021 Apr 19. PMID 33888385
- [Background] Iwata S, Ozaki M. Cerebral regional oxygen saturation as a predictive parameter for preoperative heart failure and delayed hemodynamic recovery in transcutaneous aortic valve implantation: a retrospective cohort study. J Clin Monit Comput. 2024 Aug;38(4):763-772. doi: 10.1007/s10877-024-01129-2. Epub 2024 Feb 4. PMID 38310595
- [Background] Suemori T, Horton SB, Bottrell S, Skowno JJ, Davidson A. Changes in cerebral oxygen saturation and haemoglobin concentration during paediatric cardiac surgery. Anaesth Intensive Care. 2017 Mar;45(2):220-227. doi: 10.1177/0310057X1704500212. PMID 28267944
- [Background] Uysal S, Lin HM, Trinh M, Park CH, Reich DL. Optimizing cerebral oxygenation in cardiac surgery: A randomized controlled trial examining neurocognitive and perioperative outcomes. J Thorac Cardiovasc Surg. 2020 Mar;159(3):943-953.e3. doi: 10.1016/j.jtcvs.2019.03.036. Epub 2019 Mar 29. PMID 31056357
- [Background] Parnia S, Yang J, Nguyen R, Ahn A, Zhu J, Inigo-Santiago L, Nasir A, Golder K, Ravishankar S, Bartlett P, Xu J, Pogson D, Cooke S, Walker C, Spearpoint K, Kitson D, Melody T, Chilwan M, Schoenfeld E, Richman P, Mills B, Wichtendahl N, Nolan J, Singer A, Brett S, Perkins GD, Deakin CD. Cerebral Oximetry During Cardiac Arrest: A Multicenter Study of Neurologic Outcomes and Survival. Crit Care Med. 2016 Sep;44(9):1663-74. doi: 10.1097/CCM.0000000000001723. PMID 27071068
- [Background] Heringlake M, Garbers C, Kabler JH, Anderson I, Heinze H, Schon J, Berger KU, Dibbelt L, Sievers HH, Hanke T. Preoperative cerebral oxygen saturation and clinical outcomes in cardiac surgery. Anesthesiology. 2011 Jan;114(1):58-69. doi: 10.1097/ALN.0b013e3181fef34e. PMID 21178669
- [Background] Schoen J, Meyerrose J, Paarmann H, Heringlake M, Hueppe M, Berger KU. Preoperative regional cerebral oxygen saturation is a predictor of postoperative delirium in on-pump cardiac surgery patients: a prospective observational trial. Crit Care. 2011;15(5):R218. doi: 10.1186/cc10454. Epub 2011 Sep 19. PMID 21929765
- [Background] Watzman HM, Kurth CD, Montenegro LM, Rome J, Steven JM, Nicolson SC. Arterial and venous contributions to near-infrared cerebral oximetry. Anesthesiology. 2000 Oct;93(4):947-53. doi: 10.1097/00000542-200010000-00012. PMID 11020744
- [Background] Mack MJ, Leon MB, Thourani VH, Makkar R, Kodali SK, Russo M, Kapadia SR, Malaisrie SC, Cohen DJ, Pibarot P, Leipsic J, Hahn RT, Blanke P, Williams MR, McCabe JM, Brown DL, Babaliaros V, Goldman S, Szeto WY, Genereux P, Pershad A, Pocock SJ, Alu MC, Webb JG, Smith CR; PARTNER 3 Investigators. Transcatheter Aortic-Valve Replacement with a Balloon-Expandable Valve in Low-Risk Patients. N Engl J Med. 2019 May 2;380(18):1695-1705. doi: 10.1056/NEJMoa1814052. Epub 2019 Mar 16. PMID 30883058
- [Background] Leon MB, Smith CR, Mack MJ, Makkar RR, Svensson LG, Kodali SK, Thourani VH, Tuzcu EM, Miller DC, Herrmann HC, Doshi D, Cohen DJ, Pichard AD, Kapadia S, Dewey T, Babaliaros V, Szeto WY, Williams MR, Kereiakes D, Zajarias A, Greason KL, Whisenant BK, Hodson RW, Moses JW, Trento A, Brown DL, Fearon WF, Pibarot P, Hahn RT, Jaber WA, Anderson WN, Alu MC, Webb JG; PARTNER 2 Investigators. Transcatheter or Surgical Aortic-Valve Replacement in Intermediate-Risk Patients. N Engl J Med. 2016 Apr 28;374(17):1609-20. doi: 10.1056/NEJMoa1514616. Epub 2016 Apr 2. PMID 27040324
- [Background] Leon MB, Smith CR, Mack M, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Brown DL, Block PC, Guyton RA, Pichard AD, Bavaria JE, Herrmann HC, Douglas PS, Petersen JL, Akin JJ, Anderson WN, Wang D, Pocock S; PARTNER Trial Investigators. Transcatheter aortic-valve implantation for aortic stenosis in patients who cannot undergo surgery. N Engl J Med. 2010 Oct 21;363(17):1597-607. doi: 10.1056/NEJMoa1008232. Epub 2010 Sep 22. PMID 20961243
- [Background] Vahanian A, Alfieri O, Andreotti F, Antunes MJ, Baron-Esquivias G, Baumgartner H, Borger MA, Carrel TP, De Bonis M, Evangelista A, Falk V, Lung B, Lancellotti P, Pierard L, Price S, Schafers HJ, Schuler G, Stepinska J, Swedberg K, Takkenberg J, Von Oppell UO, Windecker S, Zamorano JL, Zembala M; ESC Committee for Practice Guidelines (CPG); Joint Task Force on the Management of Valvular Heart Disease of the European Society of Cardiology (ESC); European Association for Cardio-Thoracic Surgery (EACTS). Guidelines on the management of valvular heart disease (version 2012): the Joint Task Force on the Management of Valvular Heart Disease of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS). Eur J Cardiothorac Surg. 2012 Oct;42(4):S1-44. doi: 10.1093/ejcts/ezs455. Epub 2012 Aug 25. No abstract available. PMID 22922698